CLINICAL TRIAL: NCT02786342
Title: Italian Multicentric Prospective Study Of Validation Of Angiogenesis Polymorphisms In HCC Patients Treated With Sorafenib
Brief Title: Italian Study Of Validation Of Angiogenesis Polymorphisms In HCC Patients Treated With Sorafenib
Acronym: INNOVATE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: IRSTB051
Record Dates: First submitted 2016-05-20; First posted 2016-06-01 (Estimated); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Sorafenib; HCC; Angiogenesis; Polymorphisms
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood, plasma and serum samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Advanced HCC patients treated with sorafenib
  Interventions: Procedure: blood sample collection

INTERVENTIONS:
Procedure: blood sample collection

SUMMARY:
Sorafenib represents the standard care for advanced hepatocellular carcinoma (HCC). However, molecular predictors of sorafenib efficacy have not yet been identified.

The primary aim of the study is to validate the prognostic or predictive role of eNOS,Ang2, HIF-1, VEGF and VEGFR polymorphisms in relation to clinical outcome (progression-free survival, PFS) of HCC patients treated with sorafenib.

DETAILED DESCRIPTION:
Sorafenib is a multikinase inhibitor acting on vascular endothelial growth factor receptors (VEGFR) and platelet-derived growth factor receptor beta (PDGFRβ) involved in tumor cell proliferation and tumor angiogenesis.

Angiogenesis is a cascade of linked and sequential steps ultimately leading to tumour neovascularisation. Preclinical data suggested that significant HCC growth is dependent on angiogenesis, and an increase in tumour dimension may induce vascular endothelial cell proliferation.

Vascular endothelial growth factor (VEGF)-driven pathway has been demonstrated to play a major role in tumour angiogenesis. In fact, VEGF as a potent permeability factor promotes cell migration during invasion and as an endothelial growth factor stimulates endothelial cell proliferation, inducing the budding of new blood vessels around the growing tumour masses .

Single nucleotide polymorphisms (SNPs) in VEGF and VEGF receptor (VEGFR) genes have also been correlated to tumour neoangiogenesis through different biological mechanisms.

In the ALICE-1 study HCC patients receiving sorafenib were tested for VEGF-A, VEGF-C and VEGFR-1,2,3 SNPs. At univariate analysis VEGF-A alleles C of rs25648, T of rs833061, C of rs699947, C of rs2010963, VEGF-C alleles T of rs4604006, G of rs664393, VEGFR-2 alleles C of rs2071559, C of rs2305948 were significant predictors of PFS and overall survival (OS). At multivariate analysis rs2010963, rs4604006 and Barcelona Clinic Liver Cancer (BCLC) stage resulted to be independent factors influencing PFS and OS.

In the ALICE-2 study SNPs of hypoxia inducible factor 1α (HIF-1α) were statistically significant for PFS and OS. The extended analysis of VEGF and VEGFR SNPs confirms the results of ALICE-1 study. The presence of GG genotype of rs12434438 (HIF-1α) select a population with a particularly poor outcome independently from the clinical effect of the two VEGF SNPs (PFS: 2.6 months, p<0,0001; OS: 6.6 months, p<0,0001).

In ePHAS study a training cohort of 41 HCC patients and a validation cohort of 87 patients receiving sorafenib was analyzed. At univariate analysis, patients homozygous for an endothelial nitric oxide synthase (eNOS) haplotype (HT1: T-4b at eNOS-786/eNOS VNTR) had a lower median PFS (2.6 vs. 5.8 months, p <0.0001) and OS (3.2 vs.14.6 months, p = 0.024) than those with other haplotypes. These data were confirmed in the validation set in which patients homozygous for HT1 had a lower median PFS (2.0 vs. 6.7 months, p <0.0001) and OS (6.4 vs.18.0 months, p < 0.0001).

On the basis of these premises this prospective study aims at validating the potential role of eNOS, VEGF, VEGFR, HIF-1 and Ang2 polymorphisms in patients with HCC treated with sorafenib.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent.
2. Ability to understand and the willingness to sign a written informed consent document.
3. Male or Female, aged >18 years.
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 2 or less.
5. Life expectancy of 12 weeks or more.
6. Adequate hematologic function.
7. Patients were required to have at least one untreated target lesion that could be measured in one dimension, according to the Response Evaluation Criteria in Solid Tumors (RECIST version 1.1).
8. Concomitant antiviral systemic therapy was allowed.
9. Resolution of all acute toxic effects of any prior local treatment.
10. HCC diagnosed according to the AASLD and/or EASL criteria.

Exclusion Criteria:

1. Previous or concurrent cancer that is distinct in primary site or histology from HCC.
2. Renal failure requiring hemo- or peritoneal dialysis.
3. Presence of recent (< 6 months) or current cardiac failure Known history of human immunodeficiency virus (HIV) infection.
4. Known central nervous system tumors including metastatic brain disease.
5. Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
6. Any prior local therapy within 4 weeks of study entry.
7. Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients with advanced-stage hepatocellular carcinoma, according to the criteria American Association for the Study of Liver Disease (AASLD) / European Association for the Study of the Liver (EASL)
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2016-02-15 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
PFS | up to three years
  prognostic/predictive role of eNOS,Ang2, HIF-1, VEGF and VEGFR polymorphisms in relation to Progression Free Survival

SECONDARY OUTCOMES:
OS | up to three years
  prognostic/predictive role of eNOS,Ang2, HIF-1, VEGF and VEGFR polymorphisms in relation to Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Casadei-Gardini, MD, Principal Investigator — Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST)
Locations (10):
- Italy (10):
  - IRCCS Istituto Tumori Giovanni Paolo II, Bari, BA
  - AOU di Cagliari - PO San Giovanni di Dio, Cagliari, CA
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola, FC
  - Istituto Oncologico Veneto, Padua, PD
  - Azienda Ospedaliera Universitaria Pisana, Pisa, PI
  - Oncologia medica - AOU di Parma, Parma, PR
  - Oncologia medica , PO FAENZA, Ausl della Romagna, Faenza, RA
  - Ospedale Civile degli Infermi, Rimini, RM
  - Azienda Sanitaria Universitaria Integrata di Udine S. Maria della Misericordia, Udine, UD
  - policlinico universitario Campus Bio-medico, Roma

REFERENCES:
- [Background] Llovet JM, Ricci S, Mazzaferro V, Hilgard P, Gane E, Blanc JF, de Oliveira AC, Santoro A, Raoul JL, Forner A, Schwartz M, Porta C, Zeuzem S, Bolondi L, Greten TF, Galle PR, Seitz JF, Borbath I, Haussinger D, Giannaris T, Shan M, Moscovici M, Voliotis D, Bruix J; SHARP Investigators Study Group. Sorafenib in advanced hepatocellular carcinoma. N Engl J Med. 2008 Jul 24;359(4):378-90. doi: 10.1056/NEJMoa0708857. PMID 18650514
- [Background] Scartozzi M, Faloppi L, Svegliati Baroni G, Loretelli C, Piscaglia F, Iavarone M, Toniutto P, Fava G, De Minicis S, Mandolesi A, Bianconi M, Giampieri R, Granito A, Facchetti F, Bitetto D, Marinelli S, Venerandi L, Vavassori S, Gemini S, D'Errico A, Colombo M, Bolondi L, Bearzi I, Benedetti A, Cascinu S. VEGF and VEGFR genotyping in the prediction of clinical outcome for HCC patients receiving sorafenib: the ALICE-1 study. Int J Cancer. 2014 Sep 1;135(5):1247-56. doi: 10.1002/ijc.28772. Epub 2014 Feb 20. PMID 24510746
- [Derived] Casadei-Gardini A, Marisi G, Dadduzio V, Gramantieri L, Faloppi L, Ulivi P, Foschi FG, Tamburini E, Vivaldi C, Rizzato MD, Ielasi L, Canale M, Conti F, Rudnas B, Fornaro L, Silvestris N, Silletta M, Cardellino GG, Lonardi S, Fornari F, Orsi G, Rovesti G, Zagonel V, Cascinu S, Scartozzi M. Association of NOS3 and ANGPT2 Gene Polymorphisms with Survival in Patients with Hepatocellular Carcinoma Receiving Sorafenib: Results of the Multicenter Prospective INNOVATE Study. Clin Cancer Res. 2020 Sep 1;26(17):4485-4493. doi: 10.1158/1078-0432.CCR-19-3897. Epub 2020 May 5. PMID 32371540